CLINICAL TRIAL: NCT01541423
Title: A European Multi-Center, Multi-Country, Post-Authorisation, Observational Study (Registry) Of Patients With Hereditary Angioedema (HAE) Who Are Administered CINRYZE® (C1 Inhibitor [Human]) For The Treatment Or Prevention Of HAE Attacks
Brief Title: A European Post-Authorisation Observational Study Of Patients With Hereditary Angioedema
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 0624-401; SHP616-401
Record Dates: First submitted 2012-02-16; First posted 2012-03-01 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational (non-interventional) study is being conducted to characterize the safety and use of CINRYZE in routine clinical practice when administered for (1) routine prevention of angioedema attacks, (2) pre-procedure prevention of angioedema attacks, and/or (3) treatment of angioedema attacks.

ELIGIBILITY:
Inclusion Criteria

All patients must:

* Have a diagnosis of HAE and be receiving CINRYZE for prevention or treatment of angioedema attacks
* Provide written informed consent/assent in compliance with applicable country-specific and local regulations

Exclusion Criteria

All patients must not:

* Be receiving CINRYZE in an investigational study
* Be receiving another HAE therapy as part of a clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with HAE in Europe who are receiving CINRYZE in routine clinical practice for prevention or treatment of angioedema attacks. Approximately 20 sites are planned for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2012-05-11 (Actual); Primary Completion 2016-09-25 (Actual); Study Completion 2016-09-25 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions | 12 months
Incidence of thrombotic/thromboembolic events | 12 months
Occurrence of pregnancy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (20):
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen (UZA), Antwerp, Edegem
  - Clinic St-Luc University Hospital, Brussels
- France (5):
  - CHU d'Angers, Angers
  - Hôpital Claude-Huriez, Lille
  - Immunologie Clinique et Allergologie, Nancy
  - Hôpital Saint Antoine, Paris
  - Université Paris Descartes, Paris
- Germany (6):
  - Allergie-Centrum-Charite, Berlin
  - Universitätsklinik Essen, Essen
  - Johann Wolfgang Goethe Universität, Frankfurt
  - Universität-Hautklinik Mainz, Mainz
  - Hämophilie-Zentrum Rhein Main, Mörfelden-Walldorf
  - Klinikum rechts der Isar der technischen Universität München, München
- Italy (2):
  - Ospedale Luigi Sacco, Milan
  - Azienda Ospedaliera "V. Cervello", Palermo
- Spain (3):
  - C.A.R San Pedro, Logroño
  - Hospital General Universitario, Madrid
  - Hospital Universitario La Paz, Madrid
- United Kingdom (2):
  - Barts and the London NHS Trust, London
  - Northern General Hospital, Sheffield

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fc34db2bf003ab45886